CLINICAL TRIAL: NCT00739674
Title: Randomized Open-label Trial to Evaluate the Effectiveness of Diet Management With a Losartan Titration Regimen Versus Losartan Titration Regimen Alone on Blood Pressure Reduction in Hypertensives.
Brief Title: SAALT: Subtracting Salt and Adding Losartan Trial (0954A-335)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-335; 2008_022; MK0954A-335
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Hydrochlorothiazide; Calcium Channel Blockers; Diet, Sodium-Restricted

ARMS (2):
- Losartan-Based Regimen Alone (L Group) (Active Comparator): Losartan-based regimen, with sequential titration including HCTZ and CCB as needed to achieve target blood pressure.
  Interventions: Drug: losartan potassium (+ hydrochlorothiazide [HCTZ] + calcium channel blocker [CCB])
- Diet Management and Losartan-Based Regimen (DML Group) (Experimental): Losartan with sequential titration including HCTZ and CCB as needed to achieve target blood pressure combined with low-salt intake diet.
  Interventions: Drug: losartan potassium (+ hydrochlorothiazide [HCTZ] + calcium channel blocker [CCB]); Behavioral: Low Salt Diet

INTERVENTIONS:
Drug: losartan potassium (+ hydrochlorothiazide [HCTZ] + calcium channel blocker [CCB]) — Losartan 50 mg or 100 mg once daily for 40 weeks with sequential titration including HCTZ 12.5 mg or 25 mg and CCB only as needed to achieve target blood pressure, as follows:
  Patients with mild-moderate hypertension, uncontrolled hypertension on monotherapy, or diabetes:
  * Losartan 50 mg
  * Losartan 100 mg
  * Losartan 100 mg/HCTZ 12.5 mg
  * Losartan 100 mg/HCTZ 25 mg
  * Losartan 100 mg/HCTZ 25 mg + CCB
  Patients with severe hypertension:
  * Losartan 50 mg/HCTZ 12.5 mg
  * Losartan 100 mg/HCTZ 12.5 mg
  * Losartan 100 mg/HCTZ 25 mg
  * Losartan 100 mg/HCTZ 25 mg + CCB
  * Losartan 100 mg/HCTZ 25 mg + increasing CCB
Behavioral: Low Salt Diet — Low-salt intake diet (Dietary Approaches to Stop Hypertension [DASH]) including:
  * Healthy diet
  * Reduction in sodium intake to less than 2300 mmol/day
  * Low alcohol consumption (less than 2 standard drinks/day)
  Arms: Diet Management and Losartan-Based Regimen (DML Group)

SUMMARY:
To evaluate the effectiveness of diet management with a losartan based titration regimen versus losartan based titration regimen alone on blood pressure reduction in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Non Diabetic, Newly Diagnosed And Untreated For Mild To Moderate Hypertension (blood pressure > 161; < 221; 140/90 mm Hg But < 180/110 mm Hg)
* Non diabetic, newly diagnosed and untreated for severe hypertension (blood pressure > 180/110 mm Hg but < 200/120 mm Hg); Patients who are asymptomatic with no evidence of significant end organ damage including direct pressure effects can be included. Patients in an urgency/emergency state are to be excluded
* Or Diabetic, Newly Diagnosed With Hypertension And Untreated With Mild To Moderate Hypertension (blood pressure > 161;< 221; 130/80 mm Hg But < 160/100 mm Hg); Or Patient Receiving One Antihypertensive Agent (Monotherapy Only) Used To Treat Hypertension For At Least 4 Weeks And Whose Blood Pressure Is Not Controlled: blood pressure > 161;< 221; 140/90 mm Hg But < 160/100 mm Hg Or For Diabetic And/Or Coronary Artery Disease Patients: blood pressure > 161;< 221; 130/80 mm Hg But > 161;< 221; 150/90 mm Hg
* The Antihypertensive Agent Will Need To Be Discontinued Prior To Starting Study Drug

Exclusion Criteria:

* Known Secondary Hypertension Of Any Aetiology (E.G., Uncorrected Renal Artery Stenosis, Malignant Hypertension, Hypertensive Encephalopathy. Patient With Symptomatic Heart Failure (Classes 3 And 4). Patient With A Prior Myocardial Infarction Or Stroke Within The Last 6 Months
* Patient Has Undergone Percutaneous Coronary Angioplasty, Has Had Coronary Artery Bypass Within The Last 6 Months Or Has Unstable Angina
* Patient With Anuria Or Confirmed Clinically Significant Renal Or Hepatic Dysfunction (Taken From Current/Past Medical Records) And/Or Electrolyte Imbalance Laboratory Test Within The Last 3 Months Prior To Visit 1: Serum Creatinine > 130 Ìmol/L Or Creatinine Clearance < 45 Ml/Min, Ast > 3 Times Above The Normal Range, Alt > 3 Times Above The Normal Range, Serum Potassium < 3.5 Or > 5.5 Meq/L
* Significant Liver Or Respiratory Disease, Cancer Or Other concomitant Disease That Is Likely To Affect Life Expectancy Of The Patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2009-07-01 (Actual); Study Completion 2010-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: FEB-05-2008
  Last patient out: JAN-15-2010
  Total number of sites: 109 sites in Canada
Groups:
- Losartan-Based Regimen Alone (L Group): Losartan-based regimen (50 mg or 100 mg once daily for 40 weeks) with sequential titration including hydrochlorothiazide (HCTZ) 12.5 mg or 25 mg and calcium channel blocker (CCB) as needed to achieve target blood pressure.
- Diet Management and Losartan-Based Regimen (DML Group): Losartan-based regimen (50 mg or 100 mg once daily for 40 weeks) with sequential titration including HCTZ 12.5 mg or 25 mg and CCB as needed to achieve target blood pressure combined with low-salt Dietary Approaches to Stop Hypertension (DASH) diet management.
Period: Overall Study
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Started | 535 | 457
Screening Failures | 19 | 17 (ITT population took at least one dose of the study medication and had one follow-up visit.)
Site 212 Removal | 19 (lack of source documentation & frequent discrepancies between source notes and case report entries.) | 13 (lack of source documentation & frequent discrepancies between source notes and case report entries.)
No Follow-up Data | 33 | 18
Dietician Consultation >30 Days | 1 (Patients with dietician consultations >30 days after visit 1 were not included in the data analysis.) | 9 (Patients with dietician consultations >30 days after visit 1 were not included in the data analysis.)
Intent-to-treat (ITT) Population | 463 (ITT population took at least one dose of the study medication and had one follow-up visit.) | 400 (ITT population took at least one dose of the study medication and had one follow-up visit.)
Completed | 354 | 335
Not Completed | 181 | 122
Not completed — Screening failures | 19 | 17
Not completed — Site 212 removal | 19 | 13
Not completed — No follow-up data | 33 | 18
Not completed — Dietician consultation >30 days | 1 | 9
Not completed — Adverse Event | 22 | 13
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 52 | 30
Not completed — Protocol Violation | 5 | 5
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Reason missing | 2 | 0
Not completed — Clinic closed | 6 | 4
Not completed — Patient moved | 3 | 2
Not completed — Non compliant | 4 | 0
Not completed — Unable to attend visit | 3 | 1
Not completed — Home monitoring off meds | 1 | 0
Not completed — Erectile dysfunction | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Losartan-Based Regimen Alone (L Group): Losartan-based regimen (50 mg or 100 mg once daily for 40 weeks) with sequential titration including HCTZ 12.5 mg or 25 mg and CCB as needed to achieve target blood pressure.
  The Baseline Measures are reported for the Intent-to-treat (ITT) population (i.e. took at least one dose of the study medication and returned for one follow-up visit).
- Diet Management and Losartan-Based Regimen (DML Group): Losartan-based regimen (50 mg or 100 mg once daily for 40 weeks) with sequential titration including HCTZ 12.5 mg or 25 mg and CCB as needed to achieve target blood pressure combined with low-salt DASH diet management.
  The Baseline Measures are reported for the Intent-to-treat (ITT) population (i.e. took at least one dose of the study medication and returned for one follow-up visit).
- Total: Total of all reporting groups
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group) | Total
Number analyzed (Participants) | 463 | 400 | 863
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.05 (11.54) | 54.59 (11.98) | 55.38 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 208 | 447
  Male | 224 | 192 | 416
Race/Ethnicity, Customized [Number; unit: participants]
  White | 404 | 369 | 773
  Black | 9 | 4 | 13
  Hispanic | 2 | 1 | 3
  Asian | 38 | 20 | 58
  Native Indian | 3 | 2 | 5
  Other | 7 | 4 | 11
Cardiovascular Risk [Number; unit: Participants] — Cardiovascular Risk according to Framingham Equation
  Participants
    High | 112 | 92 | 204
    Medium | 94 | 61 | 155
    Low | 218 | 216 | 434
    Not Available | 35 | 27 | 62
    Missing | 4 | 4 | 8
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 90.67 (9.19) | 91.43 (9.98) | 91.02 (9.57)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 151.23 (10.80) | 151.11 (12.55) | 151.17 (11.64)
Weight [Mean (Standard Deviation); unit: Kilograms] | 85.41 (19.95) | 89.17 (20.18) | 87.16 (20.13)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Target Blood Pressure at Week 14 From Baseline
Description: Number of Patients Achieving Target Blood Pressure (<140/90 mm Hg and <130/80 mm Hg for diabetics) from baseline after 14 weeks of treatment
Time Frame: 14 Weeks
Population: 463 and 400 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 392 and 357 patients at week 14 for L group and DML group respectively.
Measure: Number; unit: Participants
Groups:
- Losartan-Based Regimen Alone (L Group): Losartan-based regimen (50 mg or 100 mg once daily for 40 weeks) with sequential titration including HCTZ 12.5 mg or 25 mg and CCB as needed to achieve target blood pressure.
- Diet Management and Losartan-Based Regimen (DML Group): Losartan-based regimen (50 mg or 100 mg once daily for 40 weeks) with sequential titration including HCTZ 12.5 mg or 25 mg and CCB as needed to achieve target blood pressure combined with low-salt DASH diet management.
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 392 | 357
Participants
  Achieve Target Blood Pressure | 276 | 270
  Did not Achieve Target Blood Pressure | 116 | 87
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.118, Fisher Exact

2. Secondary Outcome: Number of Patients Achieving Target Blood Pressure at Week 6 From Baseline
Description: Number of Patients Achieving Target Blood Pressure (<140/90 mm Hg and <130/80 mm Hg for diabetics) from baseline after 6 weeks of treatment
Time Frame: 6 Weeks
Population: 463 and 400 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 431 and 383 patients at week 6 for L group and DML group respectively.
Measure: Number; unit: Participants
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 431 | 383
Participants
  Achieve Target Blood Pressure | 239 | 231
  Did not Achieve Target Blood Pressure | 192 | 152
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.092, Fisher Exact

3. Secondary Outcome: Number of Patients Achieving Target Blood Pressure at Week 10 From Baseline
Description: Number of Patients Achieving Target Blood Pressure (<140/90 mm Hg and <130/80 mm Hg for diabetics) from baseline after 10 weeks of treatment
Time Frame: 10 Weeks
Population: 463 and 400 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 399 and 370 patients at week 10 for L group and DML group respectively.
Measure: Number; unit: Participants
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 399 | 370
Participants
  Achieve Target Blood Pressure | 257 | 254
  Did not Achieve Target Blood Pressure | 142 | 116
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.122, Fisher Exact

4. Secondary Outcome: Number of Patients Achieving Target Blood Pressure at Week 40 From Baseline
Description: Number of Patients Achieving Target Blood Pressure (<140/90 mm Hg and <130/80 mm Hg for diabetics) from baseline after 40 weeks of treatment
Time Frame: 40 Weeks
Population: 463 and 400 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 351 and 331 patients at week 40 for L group and DML group respectively.
Measure: Number; unit: Participants
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 351 | 331
Participants
  Achieve Target Blood Pressure | 264 | 240
  Did not Achieve Target Blood Pressure | 87 | 91
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.434, Fisher Exact

5. Primary Outcome: Change in Systolic Blood Pressure From Baseline to Week 14
Time Frame: 14 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 392 | 357
mm Hg | -21.01 (14.11) | -22.74 (15.81)
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.507, Regression, Linear; Adjusted for study medication, age, gender, race, cardiovascular risk, baseline weight, and baseline waist circumference

6. Primary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 14
Time Frame: 14 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 392 | 357
mm Hg | -10.19 (9.33) | -12.05 (9.50)
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.058, Regression, Linear; [statistical method as in outcome 5, analysis 1]

7. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 6
Time Frame: 6 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 431 | 383
mm Hg | -16.81 (14.92) | -18.85 (16.18)
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.158, Regression, Linear; [statistical method as in outcome 5, analysis 1]

8. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 6
Time Frame: 6 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 431 | 383
mm Hg | -8.34 (9.29) | -9.76 (9.82)
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.064, Regression, Linear; [statistical method as in outcome 5, analysis 1]

9. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 10
Time Frame: 10 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 399 | 370
mm Hg | -19.11 (14.87) | -20.95 (16.24)
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.262, Regression, Linear; [statistical method as in outcome 5, analysis 1]

10. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 10
Time Frame: 10 Weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 399 | 370
mm Hg | -9.48 (8.80) | -11.42 (9.45)
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.026, Regression, Linear; [statistical method as in outcome 5, analysis 1]

11. Secondary Outcome: Time to Achieve the Target Blood Pressure From Baseline
Description: Time to achieve the target blood pressure (<140/90 mm Hg and <130/80 mm Hg for diabetics).
Time Frame: 14 Weeks
Population: 463 and 400 - number of patients that received at least one dose of study medication and had 1 follow-up visit (ITT population). Information available for 437 and 386 patients for L group and DML group respectively.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Number analyzed (Participants) | 437 | 386
Weeks | 7.43 [6.24 to 8.62] | 6.57 [6.29 to 6.85]
Statistical Analysis 1: Comparison: Losartan-Based Regimen Alone (L Group) vs Diet Management and Losartan-Based Regimen (DML Group); Test type: Superiority or Other; p = 0.212, Log Rank

ADVERSE EVENTS:
Description: A total of 8 patients were removed from the safety population because they did not receive at least one dose of the study medication. Therefore, the safety population was based on 984 patients (531 in the L Group and 453 in the DML Group) of the total 992 enrolled patients.
Arm/Group | Losartan-Based Regimen Alone (L Group) | Diet Management and Losartan-Based Regimen (DML Group)
Serious Adverse Events (participants affected / at risk) | 13/531 | 10/453
Other Adverse Events (participants affected / at risk) | 55/531 | 46/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Losartan-Based Regimen Alone (L Group) (N=531) | Diet Management and Losartan-Based Regimen (DML Group) (N=453)
Acute myocardial infarction (Cardiac disorders) | 0 | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 (2)
Palpitations (Cardiac disorders) | 0 | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 (1)
Tachycardia (Cardiac disorders) | 0 | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0
Inflammation (General disorders) | 0 | 1 (1)
Pseudocyst (Injury, poisoning and procedural complications) | 1 (1) | 0
Amyloidosis (Immune system disorders) | 0 | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0
Diverticulitis (Infections and infestations) | 1 (1) | 0
Gastroenteritis (Infections and infestations) | 0 | 1 (1)
Pneumonia (Infections and infestations) | 0 | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 0 | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0/0
Renal failure acute (Renal and urinary disorders) | 0 | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Hypertension (Vascular disorders) | 0 | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan-Based Regimen Alone (L Group) (N=531) | Diet Management and Losartan-Based Regimen (DML Group) (N=453)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 (1)
Arrhythmia (Cardiac disorders) | 0 | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0
Eye irritation (Eye disorders) | 1 (1) | 0
Vision blurred (Eye disorders) | 1 (1) | 0
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0
Chest pain (General disorders) | 2 (2) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0
Drug ineffective (General disorders) | 2 (2) | 0
Fatigue (General disorders) | 4 (4) | 2 (2)
Malaise (General disorders) | 1 (1) | 0
Oedema (General disorders) | 1 (2) | 0
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 0
Anal abscess (Infections and infestations) | 0 | 1 (1)
Bronchitis (Infections and infestations) | 0 | 1 (1)
Gastroenteritis (Infections and infestations) | 0 | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0
Influenza (Infections and infestations) | 1 (1) | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 (1)
Nail infection (Infections and infestations) | 0 | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 | 3 (3)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0
Wrong technique in drug usage process (Injury, poisoning and procedural complications) | 0 | 1 (1)
Blood pressure decreased (Investigations) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein abnormal (Investigations) | 1 (1) | 0
Creatinine urine increased (Investigations) | 0 | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0
Urea urine increased (Investigations) | 0 | 1 (1)
Urine output decreased (Investigations) | 0 | 1 (1)
Urine sodium increased (Investigations) | 0 | 1 (1)
Weight increased (Investigations) | 0 | 1 (1)
White blood cell count abnormal (Investigations) | 0 | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 (1)
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 11 (11) | 6 (6)
Dizziness postural (Nervous system disorders) | 0 | 1 (1)
Headache (Nervous system disorders) | 7 (8) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0
Somnolence (Nervous system disorders) | 1 (1) | 0
Syncope (Nervous system disorders) | 0 | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0
Personality disorder (Psychiatric disorders) | 0 | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 0 | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0
Erectile dysfunction (Renal and urinary disorders) | 0 | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Endometrial ablation (Surgical and medical procedures) | 0 | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 2 (2)
Labile blood pressure (Vascular disorders) | 0 | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.